CLINICAL TRIAL: NCT04131257
Title: Nurse-led Continuum of Care for People With Diabetes and Pre-diabetes in Nepal (NUCOD): Study Protocol for a Cluster Randomized Controlled Trial
Brief Title: Nurse-led Continuum of Care for People With Diabetes and Pre-diabetes in Nepal
Acronym: NUCOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Biraj Man Karmacharya, Associate Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KathmanduUSMS
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuum of care; Diabetes; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuum of care (Experimental): Trained diabetes nurses will provide continuum of care to the participants that includes: conducting community awareness campaigns, screening programs, linkage to clinical care, community follow-up counseling and support for individuals with diabetes, and prevention programs for individuals with pre-diabetes.
  Interventions: Behavioral: Nurse-led Continuum of Care
- Usual care (Active Comparator): The control group will receive usual diabetic care without the nurse coordination and supervision as in the intervention group.
  Interventions: Behavioral: Nurse-led Continuum of Care

INTERVENTIONS:
Behavioral: Nurse-led Continuum of Care — This will be a nurse-led community level prevention program for individuals with diabetes and pre-diabetes, where participants in intervention group will receive nurse-led continuum of care while control group will receive usual diabetic care.

SUMMARY:
The study aims to improve diabetes prevention, access to care and advocacy through a novel cost-effective nurse-led continuum of care approach that incorporates diabetes prevention, awareness, screening and management for low-income settings, and furthermore utilizes the endeavor to advocate for establishing standard diabetes program in Nepal.

DETAILED DESCRIPTION:
The purpose of this study will be to improve diabetes prevention, access to care and advocacy through a novel cost-effective nurse-led continuum of care approach that incorporates diabetes prevention, awareness, screening and management for low-income settings, and furthermore utilizes the endeavor to advocate for establishing standard diabetes program in Nepal.

We will conduct a two-arm, open-masked stratified cluster randomized controlled trial of a NUrse-led COntinuum of care for people with diabetes and pre-diabetes (NUCOD), with primary care centers (Outreach centers and Government health posts) as a unit of randomization. NUCOD will be delivered through the trained diabetes nurses in the community to the intervention group and the outcomes will be compared to the enhanced usual-treatment group at 6 and 12 months of the intervention. The primary outcome will be change in glycated hemoglobin (HbA1c) level among diabetes and progression to type 2 diabetes among pre-diabetes, and implementation outcomes measured using the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) framework. Outcomes will be analyzed on an intention to treat basis.

The results of this trial will provide information about the effectiveness of the NUCOD program in improving clinical outcomes for diabetes and pre-diabetes individuals, and implementation outcomes for the organization.

ELIGIBILITY:
Inclusion Criteria:

* with confirmed pre-existing type II diabetes and prediabetes at the time of our screening (i.e., pre-existing diabetes or prediabetes)
* with confirmed diagnosis of type II diabetes or prediabetes after our community screening process (i.e., newly diagnosed diabetes and prediabetes)
* is not planning to relocate outside of the current place of living in next 2 years
* is older than 18 years of age

Exclusion Criteria:

* are not psychologically capable of communication
* are diagnosed as type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1236 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) level | Baseline, 6 months, 12 months
  The HbA1c will be measured using Boronate affinity chromatography (Axis-Shield, Norway)
Change in the incidence of diabetes among individuals with pre-diabetes | 6 months, 12 months
  Electronic Health Record will be used to measure the incidence of diabetes

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline, 6 months, 12 months
  The blood pressure will be measured using mean of three measurements of systolic and diastolic blood pressure, using a Microlife automatic blood pressure measuring device
Change in lipid profile levels (HDL, LDL, Triglycerides, Total cholesterol) | Baseline, 6 months, 12 months
  LDL and HDL will be measured using the elimination method (Dialab, Austria); triglyceride using GPO-PAP (Dialab, Austria); and total cholesterol using CHOD-PAP (Dialab, Austria)
Change in Body Mass Index | Baseline, 6 months, 12 months
  Body Mass Index will be calculated as weight in kilograms divided by height in meters squared
Change in the "Reach" of people participating in the program | 6 months, 12 months
  Reach will be measured by the number of people participating in the program divided by the number of people eligible to be recruited into the program
Change in the "Adoption at the patient level" measured by the Summary of Diabetes Self-Care Activities Scale | Baseline, 6 months, 12 months
  Adoption at the patient level will be measured by the proportion of people adherent to the clinical advice in lifestyle and self-care. These will be measured by the self-reported Summary of Diabetes Self-Care Activities scale. Five areas are assessed by the scale: Diet, Exercise, Blood-glucose testing, Foot care, and Smoking status. Scale of 0-7 is used. Higher the score better is the outcome.
Change in the "Adoption at the patient level" measured by the Diabetes Treatment Satisfaction Questionnaire | Baseline, 6 months, 12 months
  The Diabetes Treatment Satisfaction Questionnaire will be used to measure patient perception of the treatment. It is composed of eight questions, each of which is scored by patients on a scale ranging from zero (e.g., "very dissatisfied", "very inconvenient") to six (e.g., "very satisfied", "very convenient"). More satisfied the patient, better is the outcome.
Change in the "Adoption at the clinic level" | 6 months, 12 months
  Adoption at the clinic level will be measured by a number of participants served using health records and examining nurses' adoption of intervention program through interviews

CONTACTS AND LOCATIONS:
Overall Officials: Biraj M Karmacharya, PhD, Principal Investigator — Kathmandu University School of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Xu DR, Dev R, Shrestha A, Zhang L, Shrestha A, Shakya P, Hughes JP, Shakya PR, Li J, Liao J, Karmacharya BM. NUrse-led COntinuum of care for people with Diabetes and prediabetes (NUCOD) in Nepal: study protocol for a cluster randomized controlled trial. Trials. 2020 May 29;21(1):442. doi: 10.1186/s13063-020-04372-5. PMID 32471476